CLINICAL TRIAL: NCT02339610
Title: Multi-Center Evaluation of Post-Operative Recovery in ATTUNE Primary, Cemented Total Knee Arthroplasty
Brief Title: Evaluation of Post-Operative Recovery in ATTUNE® Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: 13005
Record Dates: First submitted 2014-11-21; First posted 2015-01-15 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Non-inflammatory Degenerative Joint Disease
Keywords: Osteoarthritis; Post-traumatic Arthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ATTUNE Primary, Cemented Total Knee Replacement: Subjects will receive one of four available ATTUNE total knee implants:
  (CR FB, CR RP, PS FB, PS RP).
  Interventions: Device: ATTUNE Primary, Cemented Total Knee Replacement

INTERVENTIONS:
Device: ATTUNE Primary, Cemented Total Knee Replacement — Patients will undergo a primary total knee replacement using one of the four implant configurations of the ATTUNE knee ( CR FB, CR RP, PS FB, PS RP).

SUMMARY:
This post-marketing investigation will evaluate the rate of recovery of the ATTUNE knee from the time of surgery through the 6 month endpoint in patients with severely painful and/or severely disabling Non-inflammatory Degenerative Joint Disease (NIDJD).

DETAILED DESCRIPTION:
This study is designed as a prospective, multi-center, non-randomized, non-comparative, non-controlled study. A sample size of N=200 subjects will be implanted at up to 4 sites in the Netherlands. Each site is expected to implant approximately 50 Subjects (50 knees).

This study allows the participating surgeon to choose the type of ATTUNE implant they would ordinarily use in standard practice. Both resurfaced patellae and non-resurfaced patellae are permitted in this investigation; consistent with the surgeons standard of care.

Subjects will receive one of four available implants: cruciate retaining fixed bearing (CR FB), cruciate retaining rotating platform (CR RP), posterior stabilized fixed bearing (PS FB), and posterior stabilized rotating platform (PS RP).

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female and between the ages of 22 and 80 years at the time of surgery, inclusive.
* Subject was diagnosed with Non-inflammatory Degenerative Joint Disease (NIDJD).
* Subject is a suitable candidate for cemented primary total knee replacement (TKA) using the devices described in this protocol with either resurfaced or non-resurfaced patellae.
* Subject has given voluntary, written informed consent to participate in this clinical investigation and has authorized the transfer of his/her information to the study Sponsor.
* Subject is currently not bedridden
* Subject, in the opinion of the Investigator, is able to understand this clinical investigation and is willing and able to perform all study procedures and follow- up visits and co-operate with investigational procedures.
* Subject is able to speak, read, and comprehend the Informed Consent Document as well as complete the Patient Reported Outcomes Questionnaires required per the protocol in either Dutch or English translations.

Exclusion Criteria:

* The Subject is a woman who is pregnant or lactating.
* Contralateral knee has already been enrolled in this study .
* Subject had a contralateral amputation.
* Previous partial knee replacement (unicompartmental, bicompartmental or patellofemoral joint replacement), patellectomy, high tibial osteotomy or primary TKA in affected knee.
* Subject is currently experiencing radicular pain from the spine that radiates into the limb to receive TKA.
* Subject has participated in a clinical investigation with an investigational product (drug or device) in the last three months.
* Subject is currently involved in any personal injury litigation, medical-legal or worker's compensation claims.
* Subject, in the opinion of the Investigator, is a drug or alcohol abuser (in the last 5 years) or has a psychological disorder that could affect their ability to complete patient reported questionnaires or be compliant with follow-up requirements.
* Subject was diagnosed and is taking prescription medications to treat a muscular disorder that limits mobility due to severe stiffness and pain such as fibromyalgia or polymyalgia.
* Subject has a significant neurological or musculoskeletal disorder(s) or disease that may adversely affect gait or weight bearing (e.g. muscular dystrophy, multiple sclerosis, Charcot disease).
* Subject is suffering from inflammatory arthritis (e.g. rheumatoid arthritis, juvenile rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus, etc.).
* Subject has a medical condition with less than 3 years of life expectancy.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
KOOS-PS change from baseline at 6 months post-operatively, as estimated from a repeated measurements longitudinal model over all post-operative time points. | 6 Months Post-Operative minus Pre-Op
  The Knee Injury and Osteoarthritis Physical Function Short Form (KOOS-PS) will be used to measure knee function as a means of evaluating the rate of recovery.
  The (KOOS-PS) is a patient self-administered questionnaire. The questionnaire consists of 7 questions to evaluate function with activities of daily living (ADL) and higher level functioning activities (sport and recreational). Each question has 5 Likert-like response options.
  Scoring is a 0-100 point scale with 100 points considered best.

SECONDARY OUTCOMES:
KOOS-PS change from baseline of the ATTUNE knee | Pre-Op (-90 days to day of surgery), 6 weeks (1 - 60 days), 3 months (61 - 137 days), 1 year (304 - 669 days), and 2 years (670 - 913 days) post-operative
  The Knee Injury and Osteoarthritis Physical Function Short Form (KOOS-PS) will be used to measure knee function as a means of evaluating the rate of recovery.
  The (KOOS-PS) is a patient self-administered questionnaire. The questionnaire consists of 7 questions to evaluate function with activities of daily living (ADL) and higher level functioning activities (sport and recreational). Each question has 5 Likert-like response options.
  Scoring is a 0-100 point scale with 100 points considered best.
Length of Hospital Stay | Immediate-post-operative: average 1 week
  Collect days of hospitalization related to TKA procedure
Annual Survivorship | 1 year (304 - 669 days), 2 years (670 - 913 days) post-operative
  A Kaplan-Meier survival analysis will be used to calculate the survivorship of the ATTUNE implant.
Type and frequency of Adverse Events (AEs) for all enrolled subjects | Day 0 - Post-Operative Day 913
  All Serious AEs must be reported to the Sponsor per protocol. All device-related and/or procedure-related AEs must be reported to the Sponsor per protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Verdonna Huey, MS, BSN, CCRP, Study Director — DePuy Orthopaedics
Locations (4):
- Netherlands (4):
  - Rijnstate Hospital - Orthopaedic Department, Arnhem, Gelderland
  - Lievensberg Hospital Orthopaedic Department, Bergen op Zoom, North Brabant
  - Spaarne Hospital Orthopaedic Department, Hoofddorp, North Holland
  - HAGA Hospital Orthopaedic Department, The Hague, South Holland

REFERENCES:
- [Derived] van Loon C, Baas N, Huey V, Lesko J, Meermans G, Vergroesen D. Early outcomes and predictors of patient satisfaction after TKA: a prospective study of 200 cases with a contemporary cemented rotating platform implant design. J Exp Orthop. 2021 Apr 17;8(1):30. doi: 10.1186/s40634-021-00347-w. PMID 33864173